CLINICAL TRIAL: NCT06961110
Title: Evaluation of Molecular Hydrogen Supplementation to Enhance the Efficacy of Weight Loss Retreat in Overweight and Obese Adolescents. A Randomized, Double-blind, Parallel-group, Placebo-controlled Trial
Brief Title: Evaluation of Molecular Hydrogen Supplementation to Enhance the Efficacy of Weight Loss Retreat in Overweight and Obese Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Assistant professor, Palacky University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FTK_2024_110
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Body Composition; Fitness; Insulin Sensitivity; Lipid Profile; Oxidative Stress; Inflammation; Autonomic Nervous System Activity
MeSH Terms: conditions — Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular hydrogen (Experimental): Supplementation with molecular hydrogen in the form of hydrogen-rich water administered 1.5 L per day - before breakfast (500 ml), lunch (500 ml) and dinner (500 ml).
  Interventions: Dietary Supplement: Hydrogen-rich water
- Placebo (Placebo Comparator): Supplementation with drinking water administered 1.5 L per day - before breakfast (500 ml), lunch (500 ml) and dinner (500 ml).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrogen-rich water — Hydrogen-rich water with molecular hydrogen concentration 1.2-1.6 ppm. No added sugar or preservatives.
  Other Names: H2 Premium Hydrogen Water, H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Molecular hydrogen
Dietary Supplement: Placebo — Drinking water with molecular hydrogen concentration 0.0 ppm. No added sugar or preservatives.
  Other Names: H2 Premium Hydrogen Water (Placebo), H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Placebo

SUMMARY:
This randomized controlled trial evaluates whether molecular hydrogen supplementation enhances the effectiveness of a 4-week weight loss retreat in overweight and obese adolescents. Outcome measures include: body composition, physical status, blood samples (insulin sensitivity, lipid profiles, markers of oxidative stress and inflammation) and autonomic nervous system function.

DETAILED DESCRIPTION:
The aim of this randomized, double-blind, parallel-group, placebo-controlled trial is to evaluate whether molecular hydrogen supplementation enhances the effectiveness of weight loss retreat for overweight and obese adolescents. Weight loss retreat is indicated for participants based on diagnosis and recommendation of a pediatrician. During the 4-week retreat, participants follow a prescribed standardized intervention consisting of reduction diet and physical activity. The total planned number of participants is 60. Participants are randomly divided into two balanced groups, with one group receiving molecular hydrogen in the form of hydrogen-rich water and the other receiving a placebo water. The daily amount of water given (hydrogen-rich or placebo) is 1.5 L. Hydrogen-rich water is packaged in specially designed aluminum containers to minimize hydrogen leakage and ensure long-term stability with a dissolved hydrogen concentration of 1.2-1.6 ppm. Participants are unable to distinguish hydrogen-rich water from the placebo because molecular hydrogen is colorless, odorless, and tasteless. Participants monitor their physical activity, sleep, and sedentary behavior one week before to retreat and undergo baseline diagnostics (including blood sampling), three weekly interim diagnostics during retreat, and final diagnostics (including blood sampling) after four weeks. If participants are available, two follow-up diagnostics are conducted six weeks and six months after the retreat and include seven-day monitoring of physical activity, sleep, and sedentary behavior. Statistical analysis is performed at a significance level of α = 0.05 and the data is evaluated using analysis of variance. In cases of non-normality, data transformations or non-parametric alternatives are used.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index indicating overweight or obesity, as determined according to the World Health Organization's international percentile charts for children aged 5-19 years.
* Presence of a regular menstrual cycle in female participants.
* Signed informed consent from the legal representative.

Exclusion Criteria:

* High blood pressure.
* Dyslipoproteinemia.
* Cardio-respiratory disorders.
* Musculoskeletal disorders.
* Use of any medications regulating heart rhythm or the neurovegetative and hormonal system.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Body mass index | Baseline and 4 weeks
  Body mass index is calculated as the ratio of body mass (kg) to the square of body height (m2). Body mass is measured using a digital scale to the nearest 0.1 kg and body height is measured using a stadiometer to the nearest 1 cm.
Six-minute walk test | Baseline and 4 weeks
  Six-minute walk test is measured by recording the total distance the participant is able to walk on a flat surface within six minutes. The participant is instructed to walk at his/her own pace in order to walk as far as possible in the given time.

SECONDARY OUTCOMES:
Body fat | Baseline and 4 weeks
  Body fat is measured using bioelectrical impedance analysis (InBody 270, InBody, Seoul, South Korea).
30-second sit-to-stand test | Baseline and 4 weeks
  30-second sit-to-stand test is measured by counting the number of repetitions in which the participant rises from sitting in a chair and sits back down within 30 seconds.
Maximal isometric grip force | Baseline and 4 weeks
  Maximal isometric grip force is measured using a hand dynamometer. The test is performed seated, with the elbow flexed at 90 degrees, and wrist in a neutral position.
Maximal wall sit | Baseline and 4 weeks
  Maximal wall sit is measured by recording the maximum duration for which the participant can maintain a static isometric squat position against a wall.
Resting blood lactate | Baseline and 4 weeks
  The level of resting blood lactate is measured using the Lactate Scout+ (EKF Diagnostics, Cardiff, United Kingdom). Capillary blood is collected in a fasting state from the fingertip using a sterile disposable lancet. Immediately after collection, the blood sample is applied to the test strip of the lactate meter and analyzed in real time.
Homeostatic model assessment of insulin resistance | Baseline and 4 weeks
  Homeostatic model assessment of insulin resistance is calculated based on fasting glucose and fasting insulin levels measured from blood samples obtained via venipuncture by a healthcare specialist. Plasma glucose is separated by centrifugation and analyzed using an enzymatic colorimetric method. Serum insulin is separated by centrifugation and analyzed using a chemiluminescent immunoassay.
Total cholesterol | Baseline and 4 weeks
  The level of total cholesterol is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation and analyzed using an enzymatic colorimetric method.
Low-density lipoprotein | Baseline and 4 weeks
  The level of low-density lipoprotein is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation and analyzed using an enzymatic colorimetric method.
High-density lipoprotein | Baseline and 4 weeks
  The level of high-density lipoprotein is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation and analyzed using an enzymatic colorimetric method.
Triglycerides | Baseline and 4 weeks
  The level of triglycerides is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation and analyzed using an enzymatic colorimetric method.
Cortisol | Baseline and 4 weeks
  The level of cortisol is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The serum is separated by centrifugation and analyzed using a chemiluminescent immunoassay.
Fibroblast growth factor 21 | Baseline and 4 weeks
  The level of fibroblast growth factor 21 is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until ELISA analysis.
Total antioxidant capacity | Baseline and 4 weeks
  The level of total antioxidant capacity is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until analysis using the TROLOX equivalent antioxidant capacity assay.
Malondialdehydes | Baseline and 4 weeks
  The level of malondialdehydes is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until ELISA analysis.
Protein carbonyls | Baseline and 4 weeks
  The level of protein carbonyls is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until ELISA analysis.
Interleukin-6 | Baseline and 4 weeks
  The level of interleukin-6 is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until ELISA analysis.
Tumor necrosis factor alpha | Baseline and 4 weeks
  The level of tumor necrosis factor alpha is measured from a fasting blood sample obtained via venipuncture by a healthcare specialist. The plasma is separated by centrifugation, divided into cryotubes, and stored at -80°C until ELISA analysis.

OTHER OUTCOMES:
Waist circumference | Baseline and 4 weeks
  Waist circumference is be measured at the narrowest part of the torso, above the iliac crest and below the lowest rib, using a non-elastic tape.
Blood pressure | Baseline and 4 weeks
  Blood pressure is measured using a mercury sphygmomanometer.
Hydration Status | Baseline and 4 weeks
  Hydration status is assessed by measuring the urine specific gravity of morning urine sample using a refractometer (SUR-NE, ATAGO, Tokyo, Japan).
Subjective evaluation of lower limb soreness | Baseline and 4 weeks
  Subjective evaluation of lower limb soreness is measured using a Visual Analog Scale before and after a wall-sit exercise, with the duration individually adjusted to 65% of each participant's maximum hold time. The Visual Analog Scale consists of a 100 mm line ranging from 0 mm (no soreness) to 100 mm (unbearable soreness).
Heart rate variability | Baseline and 4 weeks
  Heart rate variability is measured using an ECG device (DiANS PF8, DIMEA Group, Olomouc, Czech Republic). ECG recording is performed during the orthoclinostatic maneuver in a calm room without acoustic and visual disturbances.
Physical Activity Level | Baseline and 4 weeks
  The level of physical activity is assessed using a wrist-worn tri-axial accelerometer (AX3, Axivity, Newcastle, United Kingdom). This accelerometer provides detailed data on the intensity, frequency, and duration of physical activity.
Sedentary Behavior | Baseline and 4 weeks
  Sedentary behavior is assessed using a wrist-worn tri-axial accelerometer (AX3, Axivity, Newcastle, United Kingdom). This accelerometer identifies frequency and duration of sedentary bouts.
Sleep duration | Baseline and 4 weeks
  Sleep duration and quality is assessed using a wrist-worn tri-axial accelerometer (AX3, Axivity, Newcastle, United Kingdom). This accelerometer detects sleep patterns and provides total sleep time, sleep efficiency, and the timing of sleep periods.

CONTACTS AND LOCATIONS:
Overall Officials: Darja Supikova, Principal Investigator — Palacky University, Faculty of Physical Culture
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: Beginning 1 year after the publication of results with no end date.